CLINICAL TRIAL: NCT03729778
Title: Impact of HIV-1 and Aging on Mucosal Vaccine Responses
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 16-1919
Record Dates: First submitted 2018-10-16; First posted 2018-11-05 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-06

CONDITIONS: HIV-1-infection; Human Immunodeficiency Virus; HIV/AIDS; HIV Infections
Keywords: HIV; Streptococcus pneumoniae infection; Prevnar-13; PCV-13; Pneumococcal vaccine; Pneumococcal vaccines; Streptococcus pneumoniae colonization
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Healthy control and HIV-1-infected adults aged 21-45 and 55-75 years old. For HIV-1+ undetectable plasma HIV-1 RNA and documented PPSV23. Two-time blood draw, nasopharyngeal fluid collection, physical function test, fecal collection and questionnaire. Participants will be given PCV13.
Who Masked: Participant
Masking Description: Participants with be given a screening number and a participant number as a unique identifier that does not involve their name.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV+ (Active Comparator): One time administration of Prevnar-13 vaccine to HIV+ participants
  Interventions: Biological: Prevnar-13
- HIV Negative Controls (Active Comparator): One time administration of Prevnar-13 vaccine to HIV Negative Control participants
  Interventions: Biological: Prevnar-13

INTERVENTIONS:
Biological: Prevnar-13 — One time administration of prevnar-13 vaccine

SUMMARY:
The purpose of this study is to learn more about both HIV-1 infection and advancing age, and their association with increased risk of serious infection and impaired response to the Prevnar 13 vaccine.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients will be screened to determine eligibility for the study and consented. Patients who meet eligibility requirements will be immunized with PCV 20. HIV-infected adults will be tested prior to and after vaccination by blood, nasal filter paper, and stool samples to characterize mucosal and systemic antibody responses . HIV-uninfected control adults will be tested at vaccination and post vaccination to characterize mucosal and systemic antibody responses .

ELIGIBILITY:
Inclusion Criteria:

* Veterans only (accessibility to non-veterans pending)
* Age 21-45 or 55-75 Years Old
* Have not received pneumococcal vaccine Prevnar PCV-13
* Able to attend 2-3 study visits over 1 month

HIV+:

-Undetectable Viral load

HIV negative controls:

-no history or risks for HIV infection

Exclusion Criteria:

* Spleen removed
* Chronic Kidney disease (creatinine ≥ 2.0 mg/dL)
* Active liver disease
* Currently taking: Corticosteroids (prednisone, medrol, etc), Chemotherapy, Immunosuppressive medication (cyclosporine, methotrexate, azathioprine, infliximab, adalimumab, rituximab, etanercept, etc), or illicit drugs (methamphetamine, cocaine, crack, or heroin)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine pneumococcal specific IgG levels in BAL (BronchoAlveolar Lavage) fluid and NPF (Nasopharyngeal Fluid) | A change from baseline, measured at pre-vaccination, and 1 month post vaccine
  Determine pneumococcal specific IgG levels in BAL fluid and NPF and to standardize the results we will compare it to the total levels in the BAL/NPF fluid collected at all timepoints
Determine pneumococcal specific IgG levels in serum | A change from baseline, measured at pre-vaccination, and 1 month post vaccine
  Determine pneumococcal specific IgG levels in serum 1 month post vaccination response criteria must meet >2-fold rise with a post-vaccination level >1000 ng/ml for > 7 of the 12 serotypes

CONTACTS AND LOCATIONS:
Overall Officials: Edward N Janoff, MD, Principal Investigator — University of Colorado Anschutz; Rocky Mountain Regional VAMC
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States

REFERENCES:
- [Result] Kyaw MH, Rose CE Jr, Fry AM, Singleton JA, Moore Z, Zell ER, Whitney CG; Active Bacterial Core Surveillance Program of the Emerging Infections Program Network. The influence of chronic illnesses on the incidence of invasive pneumococcal disease in adults. J Infect Dis. 2005 Aug 1;192(3):377-86. doi: 10.1086/431521. Epub 2005 Jun 23. PMID 15995950
- [Result] Nuorti JP, Whitney CG; Centers for Disease Control and Prevention (CDC). Prevention of pneumococcal disease among infants and children - use of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal polysaccharide vaccine - recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2010 Dec 10;59(RR-11):1-18. PMID 21150868
- [Result] Centers for Disease Control and Prevention (CDC). Invasive pneumococcal disease and 13-valent pneumococcal conjugate vaccine (PCV13) coverage among children aged </=59 months---selected U.S. regions, 2010--2011. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1477-81. PMID 22048728
- [Result] Bonten MJ, Huijts SM, Bolkenbaas M, Webber C, Patterson S, Gault S, van Werkhoven CH, van Deursen AM, Sanders EA, Verheij TJ, Patton M, McDonough A, Moradoghli-Haftvani A, Smith H, Mellelieu T, Pride MW, Crowther G, Schmoele-Thoma B, Scott DA, Jansen KU, Lobatto R, Oosterman B, Visser N, Caspers E, Smorenburg A, Emini EA, Gruber WC, Grobbee DE. Polysaccharide conjugate vaccine against pneumococcal pneumonia in adults. N Engl J Med. 2015 Mar 19;372(12):1114-25. doi: 10.1056/NEJMoa1408544. PMID 25785969